CLINICAL TRIAL: NCT02190812
Title: An Intelligent Evaluation of Wrist Strength for the Elderly People and Its Clinical Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201302026RINB
Record Dates: First submitted 2014-07-09; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Evaluation of Wrist Muscle Strength
Keywords: wrist muscle strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Forearm supporter (Experimental): This study measured the effect of proper forearm supporter to alleviate pain and improve the wrist and grip strength in the subjects with tennis elbow.
  Interventions: Device: Forearm supporter
- Grip ball (Experimental): In this study a portable grip ball training system is developed. This study use the grip ball to train the wrist muscle. It's expected to reduce the risk of injury of the elderly in their daily lives.
  Interventions: Device: Grip ball

INTERVENTIONS:
Device: Forearm supporter — The forearm supporter be use in tennis elbow.
  Arms: Forearm supporter
Device: Grip ball
  Arms: Grip ball

SUMMARY:
Use the system to evaluate of wrist muscle strength.

DETAILED DESCRIPTION:
The muscle strength of involved wrist muscles may be gradually reduced as aging, and impair their operating skills and even life quality of the elderly. This study has proposed an evaluation system of wrist muscle strength to grip or twist. This system consists of a torque meter (FUTEK TDF400) and three plugs/sockets for simulation of common grip or twist in daily living. This study has completed to evaluate the wrist muscle strength of men and women. In addition to the effects of age and gender, this study analyzes the influence of applied force and its plug/socket diameter on the wrist muscle strength. Simultaneously, this study measured the effect of proper forearm supporter to alleviate pain and improve the wrist and grip strength in the subjects with tennis elbow. And quantitative surface EMG was used to analyze the relationship between different forearm muscles involved. In order to achieve the user-friendly effect, this system intergraded with Cloud service and Bluetooth technology, and developed a portable and intelligent evaluation system of wrist muscle strength. It can help medical personnel to assess and analysis of real-time data. The traditional training of wrist muscle is using grip or grasp a soft tennis ball. In this study a portable grip ball training system is developed. It consists of a pressure sensor and LabVIEW program. It's expected to reduce the risk of injury of the elderly in their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 and 75 years old.
* No significant upper extremity joint pain or nerve palsy.(patients with tennis elbow typical of lateral elbow pain)
* Never received surgical treatment of upper limb joints
* No significant history of cardiovascular disease

Exclusion Criteria:

* Significant disturbance of consciousness
* Unable to communicate with hearing and speech mode
* Lack of mental ability
* Emotional instability
* Significant systemic disease
* With upper limb joints or muscles, tendons obvious lesions

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
wrist muscle strength | two years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan